CLINICAL TRIAL: NCT03902769
Title: Phase II Prospective Study to Assess Rate for Prolonged Remission With Intensive Chemotherapy in Rapid Respondents AML Patients Younger Than 61 as Demonstrated by Day 5 Examination of the First Treatment.
Brief Title: Study to Assess Length of Remission With Intensive Chemotherapy in Rapidly Responding AML Patients.
Acronym: AML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Yishai Ofran, Director of leukemia Service, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMB-250-18
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: One arm open study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No allogeneic SCT (Experimental): For standard or intermediate risk AML patients who achieved good rapid response, allogenic SCT will be excluded from treatment plan
  Interventions: Procedure: Prescribing conventional chemotherapy while with holding allo-SCT
- Standard post induction therapy (Active Comparator): For slow responding AML patients, post induction therapy will be provided according to treating physician discretion
  Interventions: Procedure: Prescribing conventional chemotherapy while with holding allo-SCT

INTERVENTIONS:
Procedure: Prescribing conventional chemotherapy while with holding allo-SCT — Prescribing conventional chemotherapy (chemotherapy consolidations or autologous SCT) while with holding allo-SCT
  Other Names: No Allogeneic for rapid responders

SUMMARY:
We previously reported results of a prospective observational study demonstrating that early response defined as reduction in bone marrow (BM) blast counts to less than 5% of BM cells by the fifth day of induction therapy is a strong predictor of remission and overall survival (Ofran Y, et al. AJH, 2015). The long term survival benefit of early response was confirmed later on after a median follow-up for surviving patients of 53 months (range 17.5-84.5).

DETAILED DESCRIPTION:
Patients diagnosed with AML, younger than 61 year of age assigned for intensive chemotherapy, and diagnosed with standard or intermediate risk AML, will undergo BM examination on the fifth day of induction. Patients in whom BM blast count at the fifth day of induction will be lower than 5% will proceed therapy with consolidations or autologous SCT with-holding the option for allo-SCT. MRD monitoring will apply to those with reliable molecular marker.

ELIGIBILITY:
Inclusion Criteria:

* AML diagnosis,
* treated with 3+7 Induction chemotherapy
* Intermediate/standard risk AML

Exclusion Criteria:

* Diagnosed of APL
* high risk molecular/cytogenetic score

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | Two years

SECONDARY OUTCOMES:
Overall survivial | two years

IPD SHARING:
Plan to Share IPD: No